CLINICAL TRIAL: NCT05886530
Title: Outcomes of Differentiated Models of Service Delivery for HIV Treatment at Sentinel Sites in South Africa (Sentinel-South Africa)
Brief Title: DSD Models at South Africa Sentinel Sites
Acronym: SENTINEL 2
Status: Active, not recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Health Economics and Epidemiology Research Office (HE2RO), University of the Witwatersrand (Unknown); Clinton Health Access Initiative, Nigeria (Other)
Responsible Party: Sponsor
Other Study IDs: H-41402; M210241 (Other: University of the Witwatersrand)
Record Dates: First submitted 2023-05-15; First posted 2023-06-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: HIV; Differentiated service delivery; South Africa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV treatment survey participants: HIV treatment patients eligible to be enrolled in the patient survey
  Interventions: Other: No intervention
- Provider survey participants: HIV treatment providers eligible to be enrolled in the provider survey
  Interventions: Other: No intervention
- Time and motion observation participants: HIV treatment providers eligible to be enrolled in the time and motion observation study
  Interventions: Other: No intervention
- HIV testing survey participants: Individuals presenting for HIV testing eligible to be enrolled in the HIV testing survey
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational data collection only.

SUMMARY:
Many countries in sub-Saharan Africa are rapidly scaling up "differentiated service delivery" (DSD) models for HIV treatment to improve the quality of care, increase access, reduce costs, and support the continued expansion and sustainability of antiretroviral therapy (ART) programs. Although there is some published evidence about the health outcomes of patients in DSD models, little is known about their impacts on healthcare providers' job satisfaction, patients' quality of life, costs to providers or patients, or how DSD models affect resource allocation at the facility level.

SENTINEL is a multi-year observational study that will collect detailed data about DSD models for ART delivery and related services from 12 healthcare facilities in Malawi, 24 in South Africa, and 12 in Zambia. The first round of SENTINEL included a patient survey, provider survey, provider time-and-motion observations, and facility resource use inventory. A survey of clients testing for HIV and a supplement to the facility resource use component to describe service delivery integration will be added for the second round. The patient survey will ask up to 10 patients enrolled in each DSD model at each study site about their experiences in HIV care and in DSD models, costs incurred seeking treatment, and preferences for HIV service delivery. The provider survey will ask up to 10 providers per site about the impact of DSD models on their positions and clinics. The time-and-motion component will directly observe the time use of a sample of providers implementing DSD models. Finally, the resource utilization component will collect facility-level data about DSD model availability and enrollment and the human and other resources needed to implement them. SENTINEL is planned to include at least four approximately annual rounds of data collection between 2021 and 2025.

As national DSD programs for HIV treatment mature, it is important to understand how individual healthcare facilities are interpreting and implementing national guidelines and how healthcare workers and clients are adapting to new models of service delivery. SENTINEL will help policy makers and program managers understand the benefits and costs of differentiated service delivery and improve resource allocation going forward.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the time and motion study are:

* Patient-facing or patient-supporting service provider at the study site (patient-supporting providers include data clerks, pharmacists, etc.)
* Directly or indirectly involved in the site's implementation of ART and DSD models
* Employed in current role at the study site for at least six months
* Provides written informed consent to participate

Inclusion criteria for provider interviews are:

* Direct or indirect service provider at the study site (indirect providers include supervisors, technical advisors, etc.)
* Directly or indirectly involved in the site's implementation of ART and DSD models
* Employed in current role at the study site for at least six months
* Provides written informed consent to participate.

Inclusion criteria for the patient survey are:

* Living with HIV and on ART for at least six months at the study site
* ≥ 18 years old (18 and older considered adult for research purposes in South Africa)
* Enrolled in a specified model of care (including conventional care) up to the target number of participants for that model and have received at least one medication refill under this model
* Provide written informed consent to participate.

Inclusion criteria for the testing survey are:

* Undergoing HIV testing at the study site or other testing site within the catchment area
* ≥ 18 years old (18 and older considered adult for research purposes in South Africa)
* Provide written informed consent to participate.

Exclusion Criteria:

Exclusion criteria for the time and motion study are:

● None.

Exclusion criteria for provider interviews are:

● None.

Exclusion criteria for the patient survey are:

* Unable to communicate in any of the languages into which the questionnaire has been translated or that is known to the research assistant
* Not physically, mentally, or emotionally able to participate in the study, in the opinion of the investigators or study staff.
* Unwilling to take the time required to complete the questionnaire on the day of consent.

Exclusion criteria for the testing survey are:

* Unable to communicate in any of the languages into which the questionnaire has been translated or that is known to the research assistant
* Not physically, mentally, or emotionally able to participate in the study, in the opinion of the investigators or study staff.
* Unwilling to take the time required to complete the questionnaire on the day of consent.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clients using the South African public health system and providers employed by that system.
Sampling Method: Non-Probability Sample
Enrollment: 15520 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient survey participants with HIV viral suppression ≤400 copies/ml at most recent test | 12 months after enrollment
  Viral suppression among ART patients enrolled and not enrolled in differentiated service delivery models

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Rosen, MPA, Principal Investigator — Department of Global Health, BU School of Public Health
Locations (1):
- Health economics and Epidemiology Research Office, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data that are collected by the study will be made available after protocol closure. Data that are owned by others (e.g. the National Department of Health) cannot be shared by the authors.
Supporting Information: Study Protocol, ICF
Time Frame: Within one year of protocol closure.

REFERENCES:
- [Derived] Mokhele I, Huber A, Rosen S, Kaiser JL, Lekodeba N, Ntjikelane V, Hendrickson C, Scott N, Pascoe S. Satisfaction with service delivery among HIV treatment clients enrolled in differentiated and conventional models of care in South Africa: a baseline survey. J Int AIDS Soc. 2024 Mar;27(3):e26233. doi: 10.1002/jia2.26233. PMID 38528370
- See also: Project website — https://sites.bu.edu/ambit/